CLINICAL TRIAL: NCT01931891
Title: Extracellular Matrix Remodeling of the Umbilical Cord and Placenta in Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Collaborators: Turgut Ozal University (Other)
Responsible Party: Principal Investigator, Ayse Kirbas, Zekai Tahir Burak Maternity and Teaching Hospital, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: ztb- wharton jelly
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-07

CONDITIONS: Alterations of ECM in Umbilical Cord ECM in Preeclampisa; Alterations of ECM in Placenta in Preeclampisa
Keywords: preeclampsia, ADAMTS , wharton jelly, extracellüler matrix, placenta
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — umbilical cord placenta
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- prreclampsia

SUMMARY:
Preeclampsia affects 2% to 8% of all pregnancies and is a major cause of maternal morbidity an mortality worldwide.Althought the primary pathology leading to preeclampsia is remain not known, complex pathophysiologic pathways and mechanisms have been described.

New blood vessels evolve during angiogenesis and vasculogenesis, two physiological processes, that play a crucial role in embryogenesis and placentation. Structural alterations in the human umbilical cord, maternal spiral arteries can cause adverse fetal consequences.Pre-eclampsia is accompanied by an extensive remodelling of the ECM of the umbilical cord. Pre-eclamptic Wharton's jelly contains higher amounts of glycosaminoglycans in comparison to control tissue.

Matrixmetalloproteinases (MMPs) are a family of proteolytic enzymes that degrade various components of the extracellular matrix (ECM). A Disintegrin And Metalloproteinases (ADAMs) and ADAMs with Thrombospondin motifs (ADAMTS) are proteinases closely related to Matrix Metalloproteinases (MMPs). Dysregulation of ADAMs and ADAMTS expression have been reported in different types of pathologies such as cancer, osteoarthritis, neurodegenerative inflammation or asthma.

The role of ADAMTS in the pathomechanism of pre-eclampsia has not been studied until now. We therefore decided to compare the ADAMTS composition of the umbilical cord and placenta from newborns of mothers with pre-eclampsia with those with normal pregnancy.

DETAILED DESCRIPTION:
Preeclampsia is a multi-systemic disorder. Despite its seriousness, the aetyology remains unknown. Current theories include abnormal placentation, cardiovascular maladaptation to pregnancy, genetic and immune mechanisms, angiogenic factors and an enhanced systemic inflammatory response. Poor placental perfusion leading to wide spread maternal endothelial dysfunction is accepted as a major mechanism.

The trophoblastic invasion of maternal vessels results many changes in extracellular matrix, which gives rise to high uteroplacental vessel distensibility to accommodate the increased blood flow. So, İn normal pregnancy, there is a wide spread vasodilatation, with increased arterial compliance and reduced peripheral vascular resistance.In preeclampsia, however, trophoblastic invasion is reduced, leading to incomplete modification of maternal spiral arteries and therefore to decreases in placental perfusion.

Pre-eclampsia is accompanied by an extensive remodelling of the ECM of the umbilical cord and placenta. Pre-eclamptic Wharton's jelly contains higher amounts of glycosaminoglycans in comparison to control tissue.

Matrix metalloproteinases (MMPs) are a family of proteolytic enzymes that degrade various components of the extracellularmatrix (ECM). These enzymes play an essential role in physiological states such as tissue remodeling, morphogenesis and wound healing anda lso in pathological processes such as tumor cell invasion and metastasis.

A Disintegrin And Metalloproteinases (ADAMs) and ADAMs with Thrombospondin motifs (ADAMTS) are proteinases closely related to Matrix Metalloproteinases (MMPs). Dysregulation of ADAMsexpression has beenreported in differenttypes of pathologies such as cancer, osteoarthritis, neurodegenerative inflammation or asthma.

Some authors suggestted that ADAM-8, -9, -10, -12, -15, -17, and ADAMTS-1 might play roles in uterus remodeling during the periimplantation period and ADAMTS-12, independent of its proteolytic activity, plays a critical role in human trophoblastic cell invasion in vitro.

Human umbilical cord is an extra-embryonic structure linking the mother and fetus during pregnancy In the umbilical cord two arteries and one vein are surrounded by a collagen-rich, myxomatous substance, called Wharton's jelly (WJ) that protect the umbilical vessels against extension, bending, twisting and compression.

The extracellular matrix (ECM) of WJ is very copious and contains significant amounts of hyaluronic acid and some sulphated glycosaminoglycans (GAGs). İts interesting that Wharton's jelly contain a low number of cells but large amounts of collagen and GAGs. Wharton's jelly plays also an important role as a storage for some compounds, such as growth factor. Previous studies demonstrated that both human umbilical cord serum and tissues contain large amounts of IGF-I and IGF-binding proteins (BPs), mainly BP-1 and BP-3.

Structural alterations in the human umbilical cord can cause adverse fetal consequences. ECM dynamics can result from changes of ECM composition, for example, because of altered synthesis or degradation of one or more ECM components, or in architecture because of altered organization. Pre-eclampsia is accompanied by an extensive remodelling of the ECM of the umbilical cord.

İt found that significant increase in collagen content in the umbilical cord arteries and vein and premature replacement of hyaluronic acid by sulfated GAGs both in the UCAs and in Wharton's jelly in preeclampsia. Pre-eclamptic Wharton's jelly contains higher amounts of glycosaminoglycans in comparison to control tissue.

The role of ADAMTS in the pathology of pre-eclampsia has not been studied until now. We therefore decided to compare the ADAMTS composition of the umbilical cord and placenta from newborns of mothers with pre-eclampsia with those with normal pregnancy.

ELIGIBILITY:
-

Inclusion Criteria:

Clinical diagnosis of preeclampsia (diagnosed per ACOG criteria)

Exclusion Criteria:

known chronic disease multipl pregnancies

Exclusion Criteria:

-

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: preeclamptic women
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-02 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
severe preclampsia | 34 weeks

CONTACTS AND LOCATIONS:
Overall Officials: ayse kirbas, md, Principal Investigator — zekai tahir burak hospital
Locations (1):
- Zekai Tahir Burak Maternity Hospital, Ankara, Turkey (Türkiye)